CLINICAL TRIAL: NCT04967859
Title: Evaluation of the Efficacy of Prophylactic Topical Gentamicin in Tunnelled Catheters for Hemodialysis: a Randomized, Double-blind Clinical Trial
Brief Title: Evaluation of the Efficacy of Prophylactic Topical Gentamicin in Tunnelled Catheters for Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Camille Pereira Caetano, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 98328718.0.0000.5411
Record Dates: First submitted 2018-11-30; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Hemodialysis Catheter Infection
Keywords: hemodialysis;; tunneled catheter; central venous catheters; infections; prevention.
MeSH Terms: conditions — Infections | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: Group 1 (control): Patients using placebo ointment in ES Group 2 (intervention): Patient using 0.1% gentamicin ointment in ES
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be allocated to two groups randomly (draw), according to the prescribed topical treatment (gentamicin or placebo). The randomization protocol will be generated by an individual other than the patients' clinical follow-up using specific software (randomization). . The randomization list as well as the identification of the bottles and the uniformity of the packages will remain under the care of the researchers who are not familiar with the patients' clinical follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (control): (Placebo Comparator): Patients using placebo ointment at the exit site of the hemodialysis catheter
  Interventions: Drug: Placebo
- Group 2 (intervention) (Experimental): Patient using 0.1% gentamicin ointment at the exit site of the hemodialysis catheter
  Interventions: Drug: 0.1% gentamicin

INTERVENTIONS:
Drug: 0.1% gentamicin — Patient using 0.1% gentamicin ointment at the exit site of the hemodialysis catheter
  Arms: Group 2 (intervention)
Drug: Placebo — Patients using placebo ointment at the exit site of the hemodialysis catheter
  Arms: Group 1 (control):

SUMMARY:
Chronic kidney disease (CKD) is a major public health problem worldwide, with a significant increase in the number of patients treated with dialysis and renal transplantation. Hemodialysis (HD) is the most widely used dialysis therapy in the world, and adequate vascular access is required. The central venous catheter (CVC), although not considered the ideal vascular access, is still widely used. Its use has a strong relation with access-related infection, whether it is an exit orifice (IES), a tunnel and the most severe, the bloodstream (BSI). Consequently CVC contributes to patients' morbidity and mortality in HD, as well as to the high cost of hemodialysis treatment.

To compare the use of 0.1% topical gentamicin with the use of placebo in the exit site (ES) of tunneled catheters in patients in chronic HD regarding the reduction in IES and BSI rates and to identify the induction of bacterial resistance to gentamicin.

DETAILED DESCRIPTION:
A randomized, double-blind clinical trial comparing the use of 0.1% gentamicin versus placebo in the ES of tunnelled catheters for hemodialysis in the prevalence and density of incidence of IES and BSI. Patients will be allocated into two groups randomly: Group 1 (control): Patients using placebo ointment in ES; Group 2 (intervention): Patient using 0.1% gentamicin ointment in ES.

ELIGIBILITY:
Inclusion criteria:

* incident and prevalent patients on hemodialysis
* Tunnelled catheter implant within 90 days of study initiation

Exclusion Criteria:

* patients under 18 years of age
* pregnant women
* other types of access for dialysis other than tunnelled catheters
* course of infection at the time of initiation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Rates of exit-site infection | 1 years
  Rates of exit-site infection (measured in events per 1,000 catheter-days)
Rates of catheter-related bloodstream infections | 1 years
  Rates of catheter-related bloodstream infections (measured in events per 1,000 catheter-days)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ponce, Study Director — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Background] Camins BC. Prevention and treatment of hemodialysis-related bloodstream infections. Semin Dial. 2013 Jul-Aug;26(4):476-81. doi: 10.1111/sdi.12117. PMID 23859190
- [Background] James MT, Conley J, Tonelli M, Manns BJ, MacRae J, Hemmelgarn BR; Alberta Kidney Disease Network. Meta-analysis: antibiotics for prophylaxis against hemodialysis catheter-related infections. Ann Intern Med. 2008 Apr 15;148(8):596-605. doi: 10.7326/0003-4819-148-8-200804150-00004. PMID 18413621
- [Background] Zacharioudakis IM, Zervou FN, Arvanitis M, Ziakas PD, Mermel LA, Mylonakis E. Antimicrobial lock solutions as a method to prevent central line-associated bloodstream infections: a meta-analysis of randomized controlled trials. Clin Infect Dis. 2014 Dec 15;59(12):1741-9. doi: 10.1093/cid/ciu671. Epub 2014 Aug 25. PMID 25156111
- [Background] Wang Y, Ivany JN, Perkovic V, Gallagher MP, Woodward M, Jardine MJ. Anticoagulants and antiplatelet agents for preventing central venous haemodialysis catheter malfunction in patients with end-stage kidney disease. Cochrane Database Syst Rev. 2016 Apr 4;4(4):CD009631. doi: 10.1002/14651858.CD009631.pub2. PMID 27039404
- [Background] Liu Y, Zhang AQ, Cao L, Xia HT, Ma JJ. Taurolidine lock solutions for the prevention of catheter-related bloodstream infections: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2013 Nov 21;8(11):e79417. doi: 10.1371/journal.pone.0079417. eCollection 2013. PMID 24278133
- [Background] Zhao Y, Li Z, Zhang L, Yang J, Yang Y, Tang Y, Fu P. Citrate versus heparin lock for hemodialysis catheters: a systematic review and meta-analysis of randomized controlled trials. Am J Kidney Dis. 2014 Mar;63(3):479-90. doi: 10.1053/j.ajkd.2013.08.016. Epub 2013 Oct 11. PMID 24125729
- [Background] Snaterse M, Ruger W, Scholte Op Reimer WJ, Lucas C. Antibiotic-based catheter lock solutions for prevention of catheter-related bloodstream infection: a systematic review of randomised controlled trials. J Hosp Infect. 2010 May;75(1):1-11. doi: 10.1016/j.jhin.2009.12.017. Epub 2010 Mar 15. PMID 20227787
- [Background] Yahav D, Rozen-Zvi B, Gafter-Gvili A, Leibovici L, Gafter U, Paul M. Antimicrobial lock solutions for the prevention of infections associated with intravascular catheters in patients undergoing hemodialysis: systematic review and meta-analysis of randomized, controlled trials. Clin Infect Dis. 2008 Jul 1;47(1):83-93. doi: 10.1086/588667. PMID 18498236
- [Background] Landry D, Braden G. Reducing catheter-related infections in hemodialysis patients. Clin J Am Soc Nephrol. 2014 Jul;9(7):1156-9. doi: 10.2215/CJN.04700514. Epub 2014 Jun 26. No abstract available. PMID 24970878